CLINICAL TRIAL: NCT05526430
Title: A Phase I Dose Escalation Study of Harmine in Healthy Subjects
Brief Title: Study of Harmine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: James Murrough (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, James Murrough, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-1458; 1R01DK128242-01A1 (NIH)
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This study will employ the continual reassessment method (CRM) to find an MTD of Harmine. It uses a statistical model to estimate the relationship between dose and DLT risk to inform decisions on dosing. It first starts with a selected target DLT rate and a mathematical model for the relationship between dose and toxicity, the prior dose-toxicity curve. After a patient experiences a DLT or not, the dose-toxicity curve is re-fit incorporating the latest outcome. The next dose assigned is that most likely to be associated with the target toxicity level (the MTD). At every step, the next patient is assigned the dose estimated to be nearest to the MTD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Harmine Dose (Experimental): There will be a total of seven possible doses that include 100 mg, 200 mg, 300 mg, 500 mg, 700 mg, 900 mg and 1200 mg. Each study subject will receive a single oral dose of harmine in this single ascending dose design.
  Interventions: Drug: Harmine Hydrochloride Capsules

INTERVENTIONS:
Drug: Harmine Hydrochloride Capsules — capsules taken orally

SUMMARY:
The present study is a phase 1 dose escalation study of harmine in healthy volunteers. The primary goal of the trial is to determine the maximum tolerated dose of harmine.

DETAILED DESCRIPTION:
The present study is a phase 1 dose escalation study of harmine in healthy volunteers. The primary goal of the trial is to determine the maximum tolerated dose of harmine. Harmine will be administered in an open-label, dose escalation design that will use the continual reassessment method to inform the next dose to test in a subject. There will be a total of seven possible doses that include 100 mg, 200 mg, 300 mg, 500 mg, 700 mg, 900 mg and 1200 mg. Each study subject will receive a single oral dose of harmine in this single ascending dose design. On the treatment day, subjects will undergo continuous medical monitoring. All adverse events will be documented and events that qualify as dose limiting toxicities (DLTs) will be used to inform dosing for the subsequent subjects.

ELIGIBILITY:
Inclusion Criteria

* Male or female aged 18-55 years;
* Participants must have a level of understanding of the English language sufficient to agree to all tests and examinations required by the study and must be able to participate fully in the informed consent process;
* Body Mass Index (BMI) between 19 and 30;
* Women of childbearing potential and men must be using an acceptable method of contraception to avoid pregnancy throughout the study as judged by the investigator;
* Women must not be breastfeeding;

Exclusion Criteria

* Children under the age of 18 and adults over the age of 55 due to concerns regarding neurodevelopmental and neurocognitive effects, respectively.
* Individuals who are underweight as defined as a BMI <19, or who are obese as defined as >30 according to the Centers for Disease Control (CDC). These criteria are in line with the goals of a phase I dose finding and pharmacokinetic study.
* Presence of a significant medical illness i.e., delirium, metastatic cancer, decompensated cardiac, liver or kidney failure, major surgery, stroke or myocardial infarction during the three months prior to entry;
* Presence of a significant neurological disease such as Parkinson's disease, primary or secondary seizure disorders, intracranial tumors, severe head trauma; neurodegenerative diseases;
* Presence of neurocognitive or dementing disorders;
* Presence or history of psychiatric disorder as diagnosed by Mini Neuropsychiatric Interview (MINI);
* Urine toxicology positive for illicit drugs or dis-allowed concomitant medications as per study protocol;
* Medications with primary central nervous system (CNS) effects are dis-allowed, including psychotropic medications, antidepressants, benzodiazepines, centrally acting hypnotic agents, and centrally acting anti-migraine therapies;
* Medications with primary cardiovascular effects are dis-allowed, including beta-adrenergic antagonists, ACE inhibitors, calcium channel blockers, and diuretics;
* Any OTC medications or herbal remedies (see concomitant medications listed above) that could interfere with the study drug, pose a risk to the subject, or contain high tyramine as outlined in the Low Tyramine Diet attachment and above in the concomitant medication summary;
* Any other medications that, in the opinion of the investigators, would pose a safety risk to the patient or that would interfere with the interpretation of study results; Positive pregnancy test at screen or on the morning of the treatment day in women of childbearing potential;
* Systolic blood pressure outside the range of 100 - 140 mmHg, diastolic blood pressure outside the range of 60 - 90 mmHg, and pulse rate at rest > 100 or < 60 bpm;
* History of positive tests for hepatitis B surface antigen, hepatitis C antibodies;
* History of HIV;
* Significant ECG abnormalities as follows:
* Heart Rate < 60 and >100 bpm
* PR Interval <120 and > 220 ms
* QRS duration < 70 and >120 ms
* QTC Interval (Bazett) > 450 ms

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Depression and Anxiety Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
As of now the study team is not plan on sharing IPD as that would not align with the approved management plan.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2022, and June 2023, a total of 34 participants signed consent with 7 failed screening.
  27 were enrolled
Groups:
- Harmine Hydrochloride 100mg; Harmine Hydrochloride 200mg; Harmine Hydrochloride 300mg; Harmine Hydrochloride 500mg: Using the CRM to inform the dose to be given to the next participant based on prior information. The CRM used a one-parameter logistic regression model to estimate the relationship between dose and dose-limiting toxicity (DLT) risk to inform decisions on dosing with a target DLT rate of 25%. It first starts with a selected target DLT rate and a mathematical model for the relationship between dose and toxicity, the prior dose-toxicity curve. After a participant experiences a DLT or not, the dose-toxicity curve is re-fit incorporating the latest outcome. At every step, the next patient is assigned the dose estimated to be nearest to the MTD. To minimize the exposure of participants to potentially toxic doses, we employed some modifications to the CRM, including starting with the lowest dose available and not skipping dose levels when escalating. Additionally, we included an early stopping rule that the study would end when either the maximum number of allowable patients treated per protocol was reached or would end early in the event that the probability of the next 10 patients being given the same dose level exceeds 90%, regardless of DLT outcomes observed.
  Each participant received a single oral dose of harmine HCl on the treatment day and was observed for 8 h with continuous medical monitoring and followed up at 24 h. Note that doses >500 mg were not used due to the stopping rule above.
Period: Overall Study
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride 300mg | Harmine Hydrochloride 500mg
Started | 10 | 12 | 4 | 1
Completed | 10 | 10 | 4 | 1
Not Completed | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Harmine 300mg and 500mg combined to maintain confidentiality of one participant in 500mg arm
Groups:
- Harmine Dose 100 mg; Harmine 200 mg; Harmine >200mg: Each study subject received a single oral dose of harmine in this single ascending dose design.
  Harmine Hydrochloride Capsules: capsules taken orally
- Total: Total of all reporting groups
Arm/Group | Harmine Dose 100 mg | Harmine 200 mg | Harmine >200mg | Total
Number analyzed (Participants) | 10 | 10 | 5 | 25
Age, Continuous [Median (Standard Deviation); unit: years] | 28.9 (6.6) | 31.1 (7.3) | 29.4 (3.9) | 29.9 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 2 | 12
  Male | 5 | 5 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 6
  Not Hispanic or Latino | 7 | 8 | 3 | 18
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 5 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 4 | 5 | 3 | 12
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 66.2 (10.8) | 69.7 (14.9) | 76 (22.6) | 69.6 (15)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.8 (2.7) | 24.5 (3.0) | 25.2 (4.0) | 24.8 (3.0)
Education level [Count of Participants; unit: Participants]
  Some college | 1 | 0 | 0 | 1
  Graduated 2-year college/trade school | 0 | 1 | 0 | 1
  Graduated 4-year college | 2 | 0 | 2 | 4
  Some graduate/professional school | 3 | 4 | 3 | 10
  Completed graduate/professional school | 4 | 5 | 0 | 9
Marital status [Count of Participants; unit: Participants]
  Married/living with someone as if married | 4 | 4 | 1 | 9
  Never married | 6 | 6 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLT which is defined if have any one of the following:
  Patient Rated Inventory of Side Effects (PRISE): 0-51, higher scores indicate more adverse events observed
  Brief Psychiatric Rating Scale (BPRS): 4 - 28, higher scores indicate more symptoms of psychosis
  Vitals: blood pressure and heart rate will all be measured - anything outside of the following ranges will be noted:
  * Symptomatic hypotension, or > 20% decrease in systolic blood pressure (SBP) from pre-dosing and an absolute SBP < 90; or
  * Symptomatic hypertension, or > 20% increase in SBP or diastolic blood pressure (DBP) from predosing and absolute SBP > 170 or DBP > 95;
  * New onset tachycardia (heart rate >100 bpm) and >20% increase from pre-dosing; or symptomatic bradycardia (heart rate <60 bpm) and > 20% decrease from pre-dosing.
  * Signs and symptoms of cardiac ischemia, defined by acute ischemic changes on ECG with or without concomitant symptoms
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride 300mg | Harmine Hydrochloride 500mg
Number analyzed (Participants) | 10 | 10 | 4 | 1
Participants | 0 | 6 | 4 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Oral Harmine HCl Based on Dose Limiting Toxicity (DLT)
Description: The MTD was determined to be between 100 and 200mg and is weight-based.
Time Frame: 24 hours
Measure: Number; unit: mg/kg
Groups:
- Harmine Hydrochloride: Each participant received a single oral dose of harmine HCl (100mg, 200mg, 300mg, or 500mg) on the treatment day and was observed for 8 h with continuous medical monitoring and followed up at 24 h.
Arm/Group | Harmine Hydrochloride
Number analyzed (Participants) | 25
mg/kg | 2.7

3. Secondary Outcome: Visual Analog Scale (VAS) - Nausea
Description: Visual Analog Scale (VAS) to characterize psychoactive effects of harmine in healthy adults. Full scale from 0-10, with higher scores indicating subjective states are experienced more strongly
Time Frame: baseline, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Harmine Hydrochloride >200mg: Using the CRM to inform the dose to be given to the next participant based on prior information. The CRM used a one-parameter logistic regression model to estimate the relationship between dose and dose-limiting toxicity (DLT) risk to inform decisions on dosing with a target DLT rate of 25%. It first starts with a selected target DLT rate and a mathematical model for the relationship between dose and toxicity, the prior dose-toxicity curve. After a participant experiences a DLT or not, the dose-toxicity curve is re-fit incorporating the latest outcome. At every step, the next patient is assigned the dose estimated to be nearest to the MTD. To minimize the exposure of participants to potentially toxic doses, we employed some modifications to the CRM, including starting with the lowest dose available and not skipping dose levels when escalating. Additionally, we included an early stopping rule that the study would end when either the maximum number of allowable patients treated per protocol was reached or would end early in the event that the probability of the next 10 patients being given the same dose level exceeds 90%, regardless of DLT outcomes observed.
  Each participant received a single oral dose of harmine HCl on the treatment day and was observed for 8 h with continuous medical monitoring and followed up at 24 h. Note that doses >500 mg were not used due to the stopping rule above.
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  baseline | 0.13 [0 to 10] | 0.33 [0 to 10] | 0.10 [0 to 10]
  0.5 hours | 0.71 [0 to 10] | 0.80 [0 to 10] | 0.12 [0 to 10]
  1 hour | 0.39 [0 to 10] | 2.40 [0 to 10] | 2.30 [0 to 10]
  1.5 hours | 0.44 [0 to 10] | 2.25 [0 to 10] | 2.82 [0 to 10]
  2 hours | 0.69 [0 to 10] | 1.78 [0 to 10] | 2.22 [0 to 10]
  3 hours | 0.25 [0 to 10] | 0.93 [0 to 10] | 1.04 [0 to 10]
  4 hours | 0.37 [0 to 10] | 0.48 [0 to 10] | 0.94 [0 to 10]
  5 hours | 0.23 [0 to 10] | 0.46 [0 to 10] | 0.60 [0 to 10]
  6 hours | 0.24 [0 to 10] | 0.29 [0 to 10] | 0.16 [0 to 10]
  7 hours | 0.28 [0 to 10] | 0.65 [0 to 10] | 0.14 [0 to 10]
  8 hours | 0.23 [0 to 10] | 0.39 [0 to 10] | 0.16 [0 to 10]
  24 hours | 0.25 [0 to 10] | 0.32 [0 to 10] | 0.08 [0 to 10]

4. Secondary Outcome: Visual Analog Scale (VAS) - Hunger
Description: as for outcome 3
Time Frame: baseline, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  baseline | 2.31 [0 to 10] | 3.91 [0 to 10] | 2.96 [0 to 10]
  0.5 hours | 4.10 [0 to 10] | 3.40 [0 to 10] | 4.32 [0 to 10]
  1 hour | 2.64 [0 to 10] | 3.58 [0 to 10] | 4.66 [0 to 10]
  1.5 hours | 5.39 [0 to 10] | 4.26 [0 to 10] | 5.88 [0 to 10]
  2 hours | 5.38 [0 to 10] | 4.74 [0 to 10] | 4.94 [0 to 10]
  3 hours | 4.68 [0 to 10] | 4.65 [0 to 10] | 5.36 [0 to 10]
  4 hours | 4.14 [0 to 10] | 4.78 [0 to 10] | 6.16 [0 to 10]
  5 hours | 2.56 [0 to 10] | 1.85 [0 to 10] | 2.54 [0 to 10]
  6 hours | 2.98 [0 to 10] | 2.02 [0 to 10] | 3.86 [0 to 10]
  7 hours | 3.66 [0 to 10] | 3.35 [0 to 10] | 4.02 [0 to 10]
  8 hours | 2.87 [0 to 10] | 4.29 [0 to 10] | 4.30 [0 to 10]
  24 hours | 3.95 [0 to 10] | 3.51 [0 to 10] | 4.74 [0 to 10]

5. Secondary Outcome: Visual Analog Scale (VAS) - Feeling High/Intoxicated
Description: as for outcome 3
Time Frame: baseline, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  baseline | 0.80 [0 to 10] | 0.44 [0 to 10] | 0.12 [0 to 10]
  0.5 hours | 0.77 [0 to 10] | 0.88 [0 to 10] | 3.52 [0 to 10]
  1 hour | 1.09 [0 to 10] | 2.23 [0 to 10] | 4.52 [0 to 10]
  1.5 hours | 1.29 [0 to 10] | 2.43 [0 to 10] | 3.1 [0 to 10]
  2 hours | 0.18 [0 to 10] | 2.27 [0 to 10] | 2.74 [0 to 10]
  3 hours | 0.54 [0 to 10] | 0.62 [0 to 10] | 0.16 [0 to 10]
  4 hours | 0.84 [0 to 10] | 0.57 [0 to 10] | 0.22 [0 to 10]
  5 hours | 0.40 [0 to 10] | 0.49 [0 to 10] | 0.22 [0 to 10]
  6 hours | 0.53 [0 to 10] | 0.66 [0 to 10] | 0.18 [0 to 10]
  7 hours | 0.76 [0 to 10] | 0.65 [0 to 10] | 0.12 [0 to 10]
  8 hours | 0.56 [0 to 10] | 0.86 [0 to 10] | 0.14 [0 to 10]
  24 hours | 0.62 [0 to 10] | 0.54 [0 to 10] | 0.12 [0 to 10]

6. Secondary Outcome: Visual Analog Scale (VAS) - Drowsiness
Description: as for outcome 3
Time Frame: baseline, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  baseline | 1.43 [0 to 10] | 2.14 [0 to 10] | 2.46 [0 to 10]
  0.5 hours | 1.98 [0 to 10] | 3.04 [0 to 10] | 3.10 [0 to 10]
  1 hour | 2.54 [0 to 10] | 3.02 [0 to 10] | 3.60 [0 to 10]
  1.5 hours | 2.58 [0 to 10] | 3.96 [0 to 10] | 4.50 [0 to 10]
  2 hours | 1.97 [0 to 10] | 3.86 [0 to 10] | 4.72 [0 to 10]
  3 hours | 1.58 [0 to 10] | 3.24 [0 to 10] | 3.46 [0 to 10]
  4 hours | 2.29 [0 to 10] | 2.56 [0 to 10] | 3.32 [0 to 10]
  5 hours | 1.10 [0 to 10] | 1.86 [0 to 10] | 2.50 [0 to 10]
  6 hours | 1.86 [0 to 10] | 1.73 [0 to 10] | 0.96 [0 to 10]
  7 hours | 1.75 [0 to 10] | 1.77 [0 to 10] | 2.92 [0 to 10]
  8 hours | 1.43 [0 to 10] | 2.20 [0 to 10] | 2.20 [0 to 10]
  24 hours | 1.80 [0 to 10] | 1.00 [0 to 10] | 2.68 [0 to 10]

7. Secondary Outcome: Visual Analog Scale (VAS) - Anxiety
Description: as for outcome 3
Time Frame: baseline, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  baseline | 0.38 [0 to 10] | 1.01 [0 to 10] | 0.42 [0 to 10]
  0.5 hours | 0.33 [0 to 10] | 0.79 [0 to 10] | 2.58 [0 to 10]
  1 hour | 1 [0 to 10] | 1.03 [0 to 10] | 1.56 [0 to 10]
  1.5 hours | 0.59 [0 to 10] | 0.76 [0 to 10] | 0.70 [0 to 10]
  2 hours | 0.53 [0 to 10] | 0.78 [0 to 10] | 0.22 [0 to 10]
  3 hours | 0.42 [0 to 10] | 0.54 [0 to 10] | 0.08 [0 to 10]
  4 hours | 0.38 [0 to 10] | 0.55 [0 to 10] | 0.28 [0 to 10]
  5 hours | 0.24 [0 to 10] | 0.58 [0 to 10] | 0.26 [0 to 10]
  6 hours | 0.28 [0 to 10] | 0.51 [0 to 10] | 0.20 [0 to 10]
  7 hours | 0.19 [0 to 10] | 0.53 [0 to 10] | 0.04 [0 to 10]
  8 hours | 0.17 [0 to 10] | 0.62 [0 to 10] | 0.12 [0 to 10]
  24 hours | 0.31 [0 to 10] | 0.57 [0 to 10] | 0.14 [0 to 10]

8. Secondary Outcome: Visual Analog Scale (VAS) - Depressed Mood
Description: as for outcome 3
Time Frame: baseline, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  baseline | 0.19 [0 to 10] | 0.33 [0 to 10] | 0.38 [0 to 10]
  0.5 hours | 1.18 [0 to 10] | 0.41 [0 to 10] | 0.16 [0 to 10]
  1 hour | 0.26 [0 to 10] | 0.28 [0 to 10] | 0.46 [0 to 10]
  1.5 hours | 0.28 [0 to 10] | 0.44 [0 to 10] | 0.24 [0 to 10]
  2 hours | 0.64 [0 to 10] | 0.38 [0 to 10] | 0.10 [0 to 10]
  3 hours | 0.22 [0 to 10] | 0.36 [0 to 10] | 0.14 [0 to 10]
  4 hours | 0.24 [0 to 10] | 0.38 [0 to 10] | 0.28 [0 to 10]
  5 hours | 0.22 [0 to 10] | 0.28 [0 to 10] | 0.84 [0 to 10]
  6 hours | 0.20 [0 to 10] | 0.18 [0 to 10] | 0.16 [0 to 10]
  7 hours | 0.31 [0 to 10] | 0.29 [0 to 10] | 0.12 [0 to 10]
  8 hours | 0.20 [0 to 10] | 0.31 [0 to 10] | 0.16 [0 to 10]
  24 hours | 0.20 [0 to 10] | 0.33 [0 to 10] | 0.12 [0 to 10]

9. Secondary Outcome: Visual Analog Scale (VAS) - Happy Mood
Description: as for outcome 3
Time Frame: baseline, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  baseline | 6.13 [0 to 10] | 5.22 [0 to 10] | 5.60 [0 to 10]
  0.5 hours | 5.73 [0 to 10] | 4.28 [0 to 10] | 5.50 [0 to 10]
  1 hour | 5.63 [0 to 10] | 4.27 [0 to 10] | 4.80 [0 to 10]
  1.5 hours | 4.90 [0 to 10] | 4.45 [0 to 10] | 3.94 [0 to 10]
  2 hours | 5.34 [0 to 10] | 3.83 [0 to 10] | 3.72 [0 to 10]
  3 hours | 5.43 [0 to 10] | 3.98 [0 to 10] | 4.12 [0 to 10]
  4 hours | 5.70 [0 to 10] | 4.50 [0 to 10] | 5.22 [0 to 10]
  5 hours | 5.10 [0 to 10] | 4.34 [0 to 10] | 4.20 [0 to 10]
  6 hours | 5.07 [0 to 10] | 4.39 [0 to 10] | 5.02 [0 to 10]
  7 hours | 5.37 [0 to 10] | 4.17 [0 to 10] | 4.32 [0 to 10]
  8 hours | 5.70 [0 to 10] | 4.19 [0 to 10] | 4.36 [0 to 10]
  24 hours | 5.84 [0 to 10] | 4.85 [0 to 10] | 4.84 [0 to 10]

10. Secondary Outcome: Visual Analog Scale (VAS) - Excitement
Description: as for outcome 3
Time Frame: baseline, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  baseline | 2.55 [0 to 10] | 2.12 [0 to 10] | 3.90 [0 to 10]
  0.5 hours | 2.35 [0 to 10] | 1.44 [0 to 10] | 3.92 [0 to 10]
  1 hour | 2.66 [0 to 10] | 2.10 [0 to 10] | 3.46 [0 to 10]
  1.5 hours | 1.53 [0 to 10] | 1.89 [0 to 10] | 2.48 [0 to 10]
  2 hours | 2.37 [0 to 10] | 2.02 [0 to 10] | 2.92 [0 to 10]
  3 hours | 2.50 [0 to 10] | 1.65 [0 to 10] | 3.16 [0 to 10]
  4 hours | 2.49 [0 to 10] | 2.29 [0 to 10] | 2.76 [0 to 10]
  5 hours | 2.25 [0 to 10] | 2.17 [0 to 10] | 2.16 [0 to 10]
  6 hours | 3.21 [0 to 10] | 1.42 [0 to 10] | 2.36 [0 to 10]
  7 hours | 2.54 [0 to 10] | 1.02 [0 to 10] | 2.68 [0 to 10]
  8 hours | 2.58 [0 to 10] | 1.39 [0 to 10] | 2.70 [0 to 10]
  24 hours | 4.01 [0 to 10] | 2.35 [0 to 10] | 2.98 [0 to 10]

11. Secondary Outcome: Visual Analog Scale (VAS) - Feeling of Control
Description: as for outcome 3
Time Frame: baseline, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  baseline | 4.00 [0 to 10] | 3.27 [0 to 10] | 3.24 [0 to 10]
  0.5 hours | 3.84 [0 to 10] | 2.00 [0 to 10] | 5.46 [0 to 10]
  1 hour | 3.14 [0 to 10] | 3.81 [0 to 10] | 3.96 [0 to 10]
  1.5 hours | 3.39 [0 to 10] | 1.91 [0 to 10] | 4.04 [0 to 10]
  2 hours | 3.48 [0 to 10] | 3.07 [0 to 10] | 4.24 [0 to 10]
  3 hours | 4.13 [0 to 10] | 2.17 [0 to 10] | 3.56 [0 to 10]
  4 hours | 4.22 [0 to 10] | 2.87 [0 to 10] | 3.56 [0 to 10]
  5 hours | 3.07 [0 to 10] | 2.51 [0 to 10] | 3.48 [0 to 10]
  6 hours | 3.75 [0 to 10] | 2.14 [0 to 10] | 4.44 [0 to 10]
  7 hours | 3.76 [0 to 10] | 1.80 [0 to 10] | 4.50 [0 to 10]
  8 hours | 3.83 [0 to 10] | 2.11 [0 to 10] | 4.56 [0 to 10]
  24 hours | 3.94 [0 to 10] | 3.52 [0 to 10] | 5.30 [0 to 10]

12. Secondary Outcome: Visual Analog Scale (VAS) - Vividness of Image
Description: as for outcome 3
Time Frame: baseline, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  baseline | 5.34 [0 to 10] | 2.99 [0 to 10] | 2.10 [0 to 10]
  0.5 hours | 5.03 [0 to 10] | 2.42 [0 to 10] | 3.50 [0 to 10]
  1 hour | 5.17 [0 to 10] | 2.94 [0 to 10] | 4.24 [0 to 10]
  1.5 hours | 5.21 [0 to 10] | 2.75 [0 to 10] | 3.76 [0 to 10]
  2 hours | 5.33 [0 to 10] | 2.57 [0 to 10] | 3.24 [0 to 10]
  3 hours | 5.82 [0 to 10] | 2.76 [0 to 10] | 2.04 [0 to 10]
  4 hours | 5.70 [0 to 10] | 2.61 [0 to 10] | 2.32 [0 to 10]
  5 hours | 5.78 [0 to 10] | 2.45 [0 to 10] | 2.02 [0 to 10]
  6 hours | 5.72 [0 to 10] | 2.21 [0 to 10] | 2.58 [0 to 10]
  7 hours | 5.70 [0 to 10] | 2.17 [0 to 10] | 2.16 [0 to 10]
  8 hours | 5.94 [0 to 10] | 2.39 [0 to 10] | 2.50 [0 to 10]
  24 hours | 5.91 [0 to 10] | 2.45 [0 to 10] | 2.20 [0 to 10]

13. Secondary Outcome: Profile of Mood States Bipolar Scale (POMS-Bi): Composed-Anxious Scale
Description: The POMS-Bi is a 72-item psychological self-report rating scale used to assess transient, distinct mood states. It is also a validated instrument for identifying the effects of drug treatments.
  Items are rated on a four-point scale from 0 "much unlike this" to 3 "much like this." It includes six bipolar scales: composed-anxious, agreeable-hostile, elated-depressed, confident-unsure, energetic-tired, and clearheaded-confused. Each subscale is scored 0-36, with higher scores associated with better mood
Time Frame: Baseline, 2, 6, 7, 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  Baseline | 33.9 [0 to 36] | 29.3 [0 to 36] | 33.6 [0 to 36]
  2 hours | 31.7 [0 to 36] | 28.5 [0 to 36] | 29 [0 to 36]
  6 hours | 31.9 [0 to 36] | 30.7 [0 to 36] | 33.6 [0 to 36]
  7 hours | 33.5 [0 to 36] | 29.1 [0 to 36] | 32.8 [0 to 36]
  8 hours | 32.7 [0 to 36] | 29.2 [0 to 36] | 31.4 [0 to 36]
  24 hours | 33.1 [0 to 36] | 29.3 [0 to 36] | 33.0 [0 to 36]

14. Secondary Outcome: Profile of Mood States Bipolar Scale (POMS-Bi): Agreeable-Hostile Scale
Description: as for outcome 13
Time Frame: Baseline, 2, 6, 7, 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  Baseline | 31.5 [0 to 36] | 28.7 [0 to 36] | 31.6 [0 to 36]
  2 hours | 30.0 [0 to 36] | 28.1 [0 to 36] | 29.2 [0 to 36]
  6 hours | 31.1 [0 to 36] | 28.1 [0 to 36] | 30.6 [0 to 36]
  7 hours | 31.8 [0 to 36] | 27.0 [0 to 36] | 30.6 [0 to 36]
  8 hours | 32.2 [0 to 36] | 27.7 [0 to 36] | 30.0 [0 to 36]
  24 hours | 33.0 [0 to 36] | 27.6 [0 to 36] | 29.8 [0 to 36]

15. Secondary Outcome: Profile of Mood States Bipolar Scale (POMS-Bi): Elated-Depression Scale
Description: as for outcome 13
Time Frame: Baseline, 2, 6, 7, 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  Baseline | 29.1 [0 to 36] | 25.6 [0 to 36] | 27.0 [0 to 36]
  2 hours | 28.1 [0 to 36] | 24.6 [0 to 36] | 24.6 [0 to 36]
  6 hours | 29.0 [0 to 36] | 25.8 [0 to 36] | 27.2 [0 to 36]
  7 hours | 28.9 [0 to 36] | 24.7 [0 to 36] | 25.6 [0 to 36]
  8 hours | 29.8 [0 to 36] | 25.0 [0 to 36] | 26.0 [0 to 36]
  24 hours | 31.4 [0 to 36] | 25.5 [0 to 36] | 26.0 [0 to 36]

16. Secondary Outcome: Profile of Mood States Bipolar Scale (POMS-Bi): Confident-Unsure Scale
Description: as for outcome 13
Time Frame: Baseline, 2, 6, 7, 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  Baseline | 27.4 [0 to 36] | 24.3 [0 to 36] | 27.4 [0 to 36]
  2 hours | 24.8 [0 to 36] | 22.6 [0 to 36] | 21.6 [0 to 36]
  6 hours | 26.5 [0 to 36] | 24.5 [0 to 36] | 22.4 [0 to 36]
  7 hours | 27.1 [0 to 36] | 22.9 [0 to 36] | 23.4 [0 to 36]
  8 hours | 27.0 [0 to 36] | 23.2 [0 to 36] | 24 [0 to 36]
  24 hours | 29.0 [0 to 36] | 24.6 [0 to 36] | 26.0 [0 to 36]

17. Secondary Outcome: Profile of Mood States Bipolar Scale (POMS-Bi): Energetic-Tired Scale
Description: as for outcome 13
Time Frame: Baseline, 2, 6, 7, 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  Baseline | 24.5 [0 to 36] | 20.9 [0 to 36] | 21.8 [0 to 36]
  2 hours | 22.0 [0 to 36] | 14.5 [0 to 36] | 7.2 [0 to 36]
  6 hours | 23.1 [0 to 36] | 20.1 [0 to 36] | 19.6 [0 to 36]
  7 hours | 23.5 [0 to 36] | 20.2 [0 to 36] | 16.2 [0 to 36]
  8 hours | 26.1 [0 to 36] | 20.5 [0 to 36] | 19.4 [0 to 36]
  24 hours | 29.3 [0 to 36] | 24.0 [0 to 36] | 20.8 [0 to 36]

18. Secondary Outcome: Profile of Mood States Bipolar Scale (POMS-Bi): Clearheaded-Confused Scale
Description: as for outcome 13
Time Frame: Baseline, 2, 6, 7, 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  Baseline | 31.1 [0 to 36] | 27.9 [0 to 36] | 31.2 [0 to 36]
  2 hours | 29.0 [0 to 36] | 24.7 [0 to 36] | 22.2 [0 to 36]
  6 hours | 30.3 [0 to 36] | 27.5 [0 to 36] | 29.6 [0 to 36]
  7 hours | 30.6 [0 to 36] | 26.9 [0 to 36] | 27.8 [0 to 36]
  8 hours | 31.2 [0 to 36] | 26.6 [0 to 36] | 28.6 [0 to 36]
  24 hours | 32.4 [0 to 36] | 28.3 [0 to 36] | 30.0 [0 to 36]

19. Secondary Outcome: Perceived Stress Scale (PSS)
Description: The PSS is a 10-item self-report scale that measures the perception of stress. Each item is rated on a scale from 0-4. Full scale from 0-40, with higher score indicating more perceived stress
Time Frame: 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  Baseline | 5.7 [0 to 40] | 7.1 [0 to 40] | 5.8 [0 to 40]
  6 hours | 6.8 [0 to 40] | 7.2 [0 to 40] | 4.8 [0 to 40]
  7 hours | 6.3 [0 to 40] | 7.8 [0 to 40] | 5.6 [0 to 40]
  8 hours | 5.7 [0 to 40] | 8.5 [0 to 40] | 5.2 [0 to 40]
  24 hours | 6.2 [0 to 40] | 7.8 [0 to 40] | 6.6 [0 to 40]

20. Secondary Outcome: Patient Rated Inventory of Side Effects (PRISE)
Description: The PRISE is a self-report Adverse Event (AE) Checklist used to qualify side effects by identifying and evaluating the tolerability of each symptom.
  Only new onset or worsening symptoms were included. Participants could report more than one AE.
Time Frame: 24 hours
Population: Participants given 300mg and 500mg were combined into one arm
Measure: Count of Participants; unit: Participants
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
Participants
  Decreased energy | 3 | 8 | 5
  Fatigue | 4 | 9 | 3
  Dizziness | 3 | 5 | 5
  Nausea/vomiting | 0 | 5 | 5
  Dizziness on standing | 1 | 3 | 5
  Poor concentration | 2 | 3 | 3
  Headache | 2 | 4 | 1
  Poor coordination | 1 | 3 | 2
  Anxiety | 1 | 1 | 2
  Restlessness | 2 | 1 | 1
  Palpitations | 1 | 2 | 1
  Dry mouth | 2 | 1 | 1
  Sleeping too much | 0 | 2 | 1
  Tremors | 0 | 3 | 0
  Blurred vision | 0 | 3 | 0
  Ringing in ears | 0 | 0 | 2
  Increased perspiration | 0 | 1 | 1
  General malaise | 0 | 1 | 0
  Difficulty sleeping | 0 | 1 | 0
  Constipation | 1 | 0 | 0

21. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)
Description: The BPRS is a 16-item clinician- administered scale that captures acute behavioral changes throughout treatment. Each item is rated on a scale from 1-7. Full scale from 16-112 with higher score indicating more worse health outcomes.
Time Frame: Baseline, 2, 6, 7, 8, and 24 hours
Population: 300mg and 500mg arm combined
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale
  Baseline | 16 [16 to 112] | 16.1 [16 to 112] | 16 [16 to 112]
  2 hours | 16 [16 to 112] | 16.3 [16 to 112] | 16 [16 to 112]
  6 hours | 16 [16 to 112] | 16 [16 to 112] | 16 [16 to 112]
  7 hours | 16 [16 to 112] | 16 [16 to 112] | 16 [16 to 112]
  8 hours | 16 [16 to 112] | 16 [16 to 112] | 16 [16 to 112]
  24 hours | 16 [16 to 112] | 16 [16 to 112] | 16 [16 to 112]

22. Secondary Outcome: Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a clinician-administered suicidal ideation and behavior rating scale used to evaluate suicide risk. Full range from 0 (low intensity suicidal ideation to 9 (high intensity suicidal ideation).
Time Frame: 24 hours
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
Number analyzed (Participants) | 10 | 10 | 5
score on a scale | 0 [0 to 9] | 0 [0 to 9] | 0 [0 to 9]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: 300mg and 500mg arm combined
Arm/Group | Harmine Hydrochloride 100mg | Harmine Hydrochloride 200mg | Harmine Hydrochloride >200mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 2/10 | 5/10 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Harmine Hydrochloride 100mg (N=10) | Harmine Hydrochloride 200mg (N=10) | Harmine Hydrochloride >200mg (N=5)
Vomiting/emesis (Gastrointestinal disorders) | 0 | 3 | 5
Dizziness (Nervous system disorders) | 2 | 1 | 1
Impaired concentration/confusion (Nervous system disorders) | 1 | 3 | 0
Drowsiness (Nervous system disorders) | 0 | 3 | 0
Visual illusion (Nervous system disorders) | 0 | 1 | 0
Auditory hallucination (Nervous system disorders) | 0 | 0 | 1
Giddiness (Nervous system disorders) | 0 | 0 | 1
Hypotension (Cardiac disorders) | 0 | 0 | 1
Vasovagal (Nervous system disorders) | 0 | 0 | 1
Tingling (Nervous system disorders) | 0 | 1 | 0
Numbness (Nervous system disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Nausea w/o vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Heaviness (General disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT05526430/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT05526430/ICF_001.pdf